CLINICAL TRIAL: NCT06062368
Title: Reducing Vertigo Associated With MRI Machines
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00413291; K23DC018302 (NIH)
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Vertigo; Dizziness
Keywords: MRI; 7 Tesla; Magnetic Vestibular Stimulation
MeSH Terms: conditions — Vertigo; Dizziness

STUDY DESIGN:
Intervention Model Description: Individuals will be randomized to one of four groups, each with a different rate of entry into and exit out of the 7 Tesla MRI machine.
Who Masked: Participant
Masking Description: The participant will be unaware of the group they are participating in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Duration (No Intervention): The participant will undergo an MRI scan using the manufacturer's rate of entry into and exit from the MRI machine. This rate of entry and exit is 20 seconds.
- 1-minute entry (Experimental): The participant will undergo an MRI scan using a slower rate of entry than that specified by the manufacturer. This rate of entry is one minute (60 seconds).
  Interventions: Behavioral: Rate of Entry
- 2-minute entry (Experimental): The participant will undergo an MRI scan using a slower rate of entry than that specified by the manufacturer. This rate of entry is two minutes (120 seconds).
  Interventions: Behavioral: Rate of Entry
- 3-minute entry (Experimental): The participant will undergo an MRI scan using a slower rate of entry than that specified by the manufacturer. This rate of entry is three minutes (180 seconds).
  Interventions: Behavioral: Rate of Entry

INTERVENTIONS:
Behavioral: Rate of Entry — The participant will enter and exit the MRI scan at a slower rate than the manufacturer entry and exit.
  Arms: 1-minute entry; 2-minute entry; 3-minute entry

SUMMARY:
Vertigo, dizziness, and imbalance are commonly reported by patients and technologists when near high-field strength magnets (>4 Tesla, T) used for magnetic resonance imaging (MRI) (1-5) Prior research from the investigators has established that the mechanism is likely a Lorentz force occurring in the inner ear, as a result of interactions with normal electrical currents in the inner ear and the strong static magnetic field of the MRI machine. The investigators have recently developed preliminary data to suggest that slower rates of entry into the magnetic field can greatly attenuate the sensations of vertigo. The explanation for this is that the rates of vestibular adaptation exceed that of the stimulus, allowed a reduction or elimination of the symptoms of vertigo. The aim of this study is to recruit individuals who are already getting an MRI scan as part of other research studies to randomize the rate of entry into and exit from the static magnetic field (i.e., before and after imaging is performed). The usual rate of entry is 20 seconds. This will be increased to one, two or three minutes. The investigators will record subjective sensations of dizziness and vertigo associated with the entry into the MRI.

DETAILED DESCRIPTION:
Vertigo and nystagmus are commonly reported in 7 Tesla MRI machines, in upwards of 2/3 of individuals. Magnetic vestibular stimulation (MVS) of the inner ear explains these symptoms. In the normal state, the inner ear has constant electric current flowing from the dark cells to the hair cells of the utricular macula through the potassium enriched endolymph. This electric current drives the utricle's exquisitely sensitive response to linear accelerations. Near the utricular macula are the cupulae of the lateral and superior semicircular canals (SCCs), which are exquisitely sensitive to angular accelerations. Inside an MRI scanner, the electric current entering the utricular macula in each ear interacts with the MRI static magnetic field to create a Lorentz (magneto-hydrodynamic (MHD) force in the endolymph that pushes on the cupulae of the nearby lateral and superior semicircular canals. The force scales linearly with magnetic field strength. Thus, when a human with an intact vestibular system lies in a 7 T MRI magnet, the Lorenz force causes the endolymph to push on the cupulae, changing activity of the angular vestibulo-ocular reflex (VOR) pathway, generating both a transient sensation of motion and a sustained beating of the eyes (nystagmus), with alternating slow phases from the VOR and quick phases that reset the position of the eye.

Adult individuals that are undergoing a 7 Tesla MRI as part of other research protocols at Kennedy-Krieger Kirby Institute, will be recruited. The usual entry into the magnetic field is a button that is pressed, that enters the magnetic field over 20 seconds, and exits the magnetic field over 20 seconds. Each participant will be randomized to one of four groups: 1) entering/exiting at the usual 20 seconds, 2) entering/exiting over 1 minute, 3) entering/exiting over 2 minutes, or 4) entering/exiting over 3 minutes. Participants will be asked to close the eyes during entry and exit. The onset of vertigo and description of the sensation will be recorded. At 15 second intervals, the participants will be asked to rate vertigo on a scale from 0 (no vertigo) to 3 (severe vertigo). The end time of vertigo sensations will also be recorded. The same procedure will be completed when exiting the MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will be undergoing an MRI scan at a 7 Tesla MRI.

Exclusion Criteria:

* Exclusion criteria include pacemaker, defibrillator wires, metal implants, cochlear implants, or ferromagnetic surgical clips in the brain.
* Pregnancy
* Claustrophobia occurs in perhaps 5% of patients, and they will not proceed with the test. All subjects will fill out the routine pretesting MRI questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of vertigo symptoms | During MRI up to 6 minutes
  Participants will report the presence and intensity of their vertigo. The presence or absence of vertigo for each group will be the primary outcome.

SECONDARY OUTCOMES:
Intensity of Vertigo | During MRI up to 6 minutes
  Participants will report the intensity of their vertigo symptoms when entering and exiting the MRI scan on a scale from 0 (no vertigo)-3 (severe vertigo) at 15 second intervals. 0=no vertigo, 1=mild vertigo, 2=moderate vertigo, 3=severe vertigo
Duration (seconds) of Vertigo | During MRI up to 6 minutes
  Participants will report the onset and cessation of their vertigo symptoms when entering and exiting the MRI scanner. The duration will be calculated in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Ward, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be used only by the investigators participating in this study at Johns Hopkins University School of Medicine.

REFERENCES:
- [Background] Mian OS, Li Y, Antunes A, Glover PM, Day BL. Effect of head pitch and roll orientations on magnetically induced vertigo. J Physiol. 2016 Feb 15;594(4):1051-67. doi: 10.1113/JP271513. Epub 2015 Dec 30. PMID 26614577
- [Background] Mian OS, Li Y, Antunes A, Glover PM, Day BL. On the vertigo due to static magnetic fields. PLoS One. 2013 Oct 30;8(10):e78748. doi: 10.1371/journal.pone.0078748. eCollection 2013. PMID 24205304
- [Background] Roberts DC, Marcelli V, Gillen JS, Carey JP, Della Santina CC, Zee DS. MRI magnetic field stimulates rotational sensors of the brain. Curr Biol. 2011 Oct 11;21(19):1635-40. doi: 10.1016/j.cub.2011.08.029. Epub 2011 Sep 22. PMID 21945276
- [Result] Ward BK, Roberts DC, Otero-Millan J, Zee DS. A decade of magnetic vestibular stimulation: from serendipity to physics to the clinic. J Neurophysiol. 2019 Jun 1;121(6):2013-2019. doi: 10.1152/jn.00873.2018. Epub 2019 Apr 10. PMID 30969883